CLINICAL TRIAL: NCT01607164
Title: Depression Prevention and Management Project
Brief Title: Healthy Mood Internet Recruitment Study
Acronym: DPC-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DPC-R; 1R34MH091231-01 (NIH)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Recruitment
Keywords: Mood management; self-help; depression; prevention; cognitive behavioral
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Online self-help mood management (Experimental): Healthy Mood Project Website
  Online self-help automated mood management course available in Spanish and English via a website.
  Intervention consisted of 8 cognitive-behavioral mood management lessons.
  Interventions: Behavioral: Healthy Mood Project Website

INTERVENTIONS:
Behavioral: Healthy Mood Project Website — Self-help automated online mood management course based on cognitive-behavioral methods to control depressed mood.
  Other Names: Self-help automated Website

SUMMARY:
This study is pilot testing a self-help automated Website (similar to a self-help book) designed to help individuals to learn methods to manage their mood. The methods are cognitive-behavioral skills found effective in the treatment of depression when provided by live therapists. The purpose of the study is to determine the number of individuals who will visit the site, use the site, and respond to online surveys reporting their mood levels while using the site, and at 1, 3, and 6 months after starting to use the site. The investigators want to eventually examine whether learning these methods online would help prevent depression.

DETAILED DESCRIPTION:
Self-help automated website in Spanish and English consisting of an 8-lesson course on mood management based on cognitive behavioral methods.

Accessible via the web.

Follow-up assessments conducted at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* valid email address
* fluent in English

Exclusion Criteria:

* less than 18 years of age
* no valid email address
* not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1226 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Recruitment | One year
  Number of participants enrolling in the site per month

SECONDARY OUTCOMES:
PHQ-9 | Screening, plus 1, 3, and 6 months later
  Depression symptom measure

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Muñoz, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psychiatry at San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Munoz RF, Beardslee WR, Leykin Y. Major depression can be prevented. Am Psychol. 2012 May-Jun;67(4):285-95. doi: 10.1037/a0027666. PMID 22583342